CLINICAL TRIAL: NCT06488131
Title: A Comparative Study Between MTA Pulpotomy and Root Canal Treatment in Management of First Permanent Molars With Irreversible Pulpitis in Children: A Randomized Controlled Trial
Brief Title: Comparing MTA Pulpotomy to Root Canal Treatment in Management of Permanent Molars With Irreversible Pulpitis in Children
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alaa Eissa, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED2024-D2
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Irreversible Pulpitis
Keywords: Endodontic Treatment, Vital Pulp Therapy
MeSH Terms: interventions — Endodontics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA Pulpotomy (Experimental): Local anesthesia for pain control will be administered, followed by rubber dam isolation. Then, the tooth and surrounding rubber dam will be flushed with chlorhexidine solution for disinfection. After caries removal, a sterile bur will be used for access opening and complete deroofing of the pulp chamber. Coronal pulp tissue will be removed to the level of canal orifices using a sterile, sharp spoon excavator. A cotton pellet dampened with sodium hypochlorite will be applied on canal orifices to achieve hemostasis. This will be followed by MTA application and glass ionomer restoration. If necessary, the tooth will be restored with stainless steel crown after one week.
  Interventions: Procedure: MTA Pulpotomy
- Root Canal Treatment (Active Comparator): Local anesthesia for pain control will be administered, followed by rubber dam isolation. Then, the tooth and surrounding rubber dam will be flushed with chlorhexidine solution for disinfection. After caries removal, a sterile bur will be used for access opening and complete deroofing of the pulp chamber. Length of the root canal will be obtained using an apex locator. This will be followed by mechanical shaping using files, and irrigation with 2.5 percent sodium hypochlorite, followed by drying of the canals using paper points. Obturation will then be accomplished using gutta percha and sealer. Finally, the tooth will be restored with conventional glass ionomer restoration. If necessary, the tooth will be restored with stainless steel crown after one week.
  Interventions: Procedure: Root Canal Treatment

INTERVENTIONS:
Procedure: MTA Pulpotomy — Complete coronal MTA pulpotomy.
  Other Names: Vital Pulp Therapy
  Arms: MTA Pulpotomy
Procedure: Root Canal Treatment — Conventional root canal treatment.
  Other Names: Endodontic Treatment
  Arms: Root Canal Treatment

SUMMARY:
Dental caries, highly prevalent amongst children, can cause pulpitis. Coronal pulpotomy provides an easier, cost-effective, conservative and biologically-driven treatment option compared to endodontic treatment in mature permanent teeth with irreversible pulpitis.

The aim of the current study is to evaluate postoperative pain, clinical and radiographic outcomes of MTA pulpotomy compared to root canal treatment in children's first permanent molars suffering from irreversible pulpitis.

DETAILED DESCRIPTION:
In this randomized controlled trial, patients aged 10-14 years suffering from irreversible pulpitis in the first permanent molar with closed apex will be randomly divided into two groups. The first group will receive complete coronal MTA pulpotomy, while the second group will receive endodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children, aged 10 to 14 years
* Signs and symptoms of irreversible pulpitis in carious first permanent molar.

Exclusion Criteria:

* Molars with immature roots
* Non-restorable molars, with abnormal mobility or increased probing pocket depth (normal range = 1-3 mm)
* Any indication of pulpal necrosis, such as sinus tract or swelling or no bleeding from orifices after access opening.
* Any signs of periapical or furcal rarefaction.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pain Relief | preoperatively, immediately postoperatively and every 24 hours for 7 days after the first appointment.
  A 10 cm visual analogue scale will be used to record pain

SECONDARY OUTCOMES:
Clinical Evaluation | 3, 6, 12 and 18 months postoperatively
  * Absence of pain or discomfort
  * Tooth is functional, with no tenderness to palpation or percussion
  * Normal mobility and probing depth
  * Soft tissues surrounding the tooth are normal, with no swelling or inflammation
Radiographic Evaluation | 6, 12 and 18 months postoperatively
  * No evident radiographic periapical or furcal pathosis
  * No evident root resorption
  * Normal lamina dura

CONTACTS AND LOCATIONS:
Overall Officials: Alaa A. Eissa, Msc, Principal Investigator — Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement.

REFERENCES:
- [Result] Galani M, Tewari S, Sangwan P, Mittal S, Kumar V, Duhan J. Comparative Evaluation of Postoperative Pain and Success Rate after Pulpotomy and Root Canal Treatment in Cariously Exposed Mature Permanent Molars: A Randomized Controlled Trial. J Endod. 2017 Dec;43(12):1953-1962. doi: 10.1016/j.joen.2017.08.007. Epub 2017 Oct 20. PMID 29061359
- [Result] Taha NA, Abuzaid AM, Khader YS. A Randomized Controlled Clinical Trial of Pulpotomy versus Root Canal Therapy in Mature Teeth with Irreversible Pulpitis: Outcome, Quality of Life, and Patients' Satisfaction. J Endod. 2023 Jun;49(6):624-631.e2. doi: 10.1016/j.joen.2023.04.001. Epub 2023 Apr 19. PMID 37080387
- [Result] Asgary S, Eghbal MJ, Shahravan A, Saberi E, Baghban AA, Parhizkar A. Outcomes of root canal therapy or full pulpotomy using two endodontic biomaterials in mature permanent teeth: a randomized controlled trial. Clin Oral Investig. 2022 Mar;26(3):3287-3297. doi: 10.1007/s00784-021-04310-y. Epub 2021 Dec 2. PMID 34854987
- [Result] Beauquis J, Setbon HM, Dassargues C, Carsin P, Aryanpour S, Van Nieuwenhuysen JP, Leprince JG. Short-Term Pain Evolution and Treatment Success of Pulpotomy as Irreversible Pulpitis Permanent Treatment: A Non-Randomized Clinical Study. J Clin Med. 2022 Jan 31;11(3):787. doi: 10.3390/jcm11030787. PMID 35160239